CLINICAL TRIAL: NCT04826120
Title: Continuous Versus Intermittent Administration of Epidural Analgesia During Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor, head of department of anesthesia and critical care, Mongi Slim Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Epidural in Labor
Record Dates: First submitted 2021-03-26; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Epidural; Analgesia
Keywords: Epidural, Analgesia, Labor, delivery
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: parturients randomized in 2 groups and receiving 2 different interventions
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCEA group (Active Comparator): Patients of this group had intermittent epidural analgesia via PCEA associated to systematic 8 ml boluses every 60 min during the second stage of labor.
  Interventions: Procedure: PCEA Infusion
- CEI Group (Experimental): Patients of this group had continuous epidural infusion at the rate of 8 ml/h during the second stage of labor.
  Interventions: Procedure: Continuous epidural infusion

INTERVENTIONS:
Procedure: PCEA Infusion — Patients of this group Had PCEA during the second stage of labor
  Arms: PCEA group
Procedure: Continuous epidural infusion — Patients of this group Had continuous epidural infusion during the second stage of labor
  Arms: CEI Group

SUMMARY:
prospective randomized single blind study, including full term adult parturients, ASA 2, 3 status, scheduled for vaginal delivery. patients were randomized at 3 cm of cervix dilatation, into 2 groups.

Epidural analgesia was initiated and maintained with a solution of Bupivacaine 0,125% and Sufentanil 0,25 mcg/ml. After an initial bolus of 16 ML, patients were randomly assigned to receive intermittent boluses of 8 ml every 60 minutes after the initial dose followed by supplementary PCEA boluses of 8 ml for the first group ( PCEA group) or a continuous epidural infusion at the rate of 8 ml/h adjustable and starting immediately after The initial bolus of 16 ml for patients of the second group (CEI Group).

DETAILED DESCRIPTION:
prospective randomized single blind study, including full term adult parturients, ASA 2, 3 status, scheduled for vaginal delivery. patients were randomized at 3 cm of cervix dilatation, into 2 groups.

Epidural analgesia was initiated and maintained with a solution of Bupivacaine 0,125% and Sufentanil 0,25 mcg/ml. After an initial bolus of 16 ML, patients were randomly assigned to receive intermittent boluses of 8 ml every 60 minutes after the initial dose followed by supplementary PCEA boluses of 8 ml for the first group ( PCEA group) or a continuous epidural infusion at the rate of 8 ml/h adjustable and starting immediately after The initial bolus of 16 ml for patients of the second group (CEI Group).

The main outcome of this study was: the incidence of motor Blockage. Our secondary outcomes were: maternal satisfaction, local anaesthetic and sufentanil cumulated doses, duration of the second stage of labor, mode of delivery and pain during labor using the Visual analogic score (VAS score).

ELIGIBILITY:
Inclusion Criteria:

* Full term parturients scheduled for vaginal delivery

Exclusion Criteria:

* patients in whom cesarean section delivery was indicated during labor

Min Age: 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — parturients scheduled for vaginal delivery
Enrollment: 54 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of motor Blockage | during the epidural analgesia
  Bromage scale 1, 2 or 3

CONTACTS AND LOCATIONS:
Locations (2):
- Tunisia (2):
  - Mongi Slim University Hospital, La Marsa, Tunis Governorate
  - Mongi Slim Hospital, Tunis

IPD SHARING:
Plan to Share IPD: No